CLINICAL TRIAL: NCT04836637
Title: ValoRization of Dairy Sidestreams to Fight Calcium dEficits iN Postmenopausal Women - A Randomized Controlled Double-blinded Intervention Trial
Brief Title: ValoRization of Dairy Sidestreams to Fight Calcium dEficits iN Postmenopausal Women
Acronym: RENEW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Zealand University Hospital (Other)
Responsible Party: Principal Investigator, Inge Tetens, Professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: M236
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — maltodextrin; Calcium Carbonate; Inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Product with placebo (no calcium supplementation). (Placebo Comparator): Maltodextrin with 0 mg calcium in capsules and sachets consumed orally daily for one year.
  Interventions: Dietary Supplement: Maltodextrin
- Product with calcium-carbonate (Active Comparator): 800 mg calcium as calcium-carbonate in capsules and sachets consumed orally daily for one year.
  Interventions: Dietary Supplement: Calcium-carbonate
- Product with calcium-enriched permeate "Capolac" (Experimental): 800 mg of calcium from calcium-enriched permeate in capsules and sachets consumed orally daily for one year.
  Interventions: Dietary Supplement: Calcium-enriched permeate
- Product with calcium-enriched permeate "Capolac" and Inulin (Experimental): 800 mg of calcium from calcium-enriched permeate and 12 g inulin in capsules and sachets consumed orally daily for one year.
  Interventions: Dietary Supplement: Calcium-enriched permeate with Inulin

INTERVENTIONS:
Dietary Supplement: Maltodextrin — Three capsules are to be consumed with one sachet dissolved in 200 ml. of water for breakfast and later for dinner resulting in a total of six capsules and two sachets via oral consumption daily.
  Arms: Product with placebo (no calcium supplementation).
Dietary Supplement: Calcium-carbonate — Three capsules are to be consumed with one sachet dissolved in 200 ml. of water for breakfast and later for dinner resulting in a total of six capsules and two sachets via oral consumption daily.
  Arms: Product with calcium-carbonate
Dietary Supplement: Calcium-enriched permeate — Three capsules are to be consumed with one sachet dissolved in 200 ml. of water for breakfast and later for dinner resulting in a total of six capsules and two sachets via oral consumption daily.
  Other Names: Capolac
  Arms: Product with calcium-enriched permeate "Capolac"
Dietary Supplement: Calcium-enriched permeate with Inulin — Three capsules are to be consumed with one sachet dissolved in 200 ml. of water for breakfast and later for dinner resulting in a total of six capsules and two sachets via oral consumption daily.
  Other Names: Capolac Inulin
  Arms: Product with calcium-enriched permeate "Capolac" and Inulin

SUMMARY:
The primary objective of this study is to investigate the effects of 12-months supplementation with calcium-enriched permeate, taken alone or in conjunction with inulin, on changes in markers of bone formation and resorption and in bone mass density (BMD) in apparently healthy postmenopausal women compared with calcium-carbonate or maltodextrin supplementation.

DETAILED DESCRIPTION:
The study will include an information visit, a randomization visit, a month 3 visit and a final visit at month 12. Besides, two visits at month 6 and 9 for dispensing of trial products. Outcome parameters will be measured using blood samples obtained at the randomization visit, the month 3 visit and at the final visit at month 12. Outcome parameters will moreover be analyzed based on DXA scan obtained at the randomization visit and at the final visit at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Subject is between 45 years and 65 years of age by the time of inclusion.
* Subject has been menopausal for at least 1 year, defined as 12 months after last bleeding and up to 10 years.
* Subject is Caucasian.
* Has a BMI below 35.0.
* Holder of a computer.
* Has a sufficient vitamin D status (plasma 25OHD concentration > 50 nmol/L).
* Subject is willing and able to provide written informed consent prior to participation.

Exclusion Criteria:

* Subject taking supplements or medicine that affects calcium and bone metabolism e.g. diuretics or hormone replacement therapy evaluated by the investigator.
* Intake of antibiotics in the last 3 months before enrollment.
* Subject with an osteoporosis diagnosis or history of osteoporotic fractures.
* Presence of renal, gastrointestinal, hepatic or endocrinological diseases.
* Subject with any serious illness or history of cancer within the past 5 years (except adequately-treated localized basal cell skin cancer or in situ uterine cervical cancer).
* Known or suspected abuse of alcohol or recreational drugs.
* Known milk allergy.
* Known or suspected hypersensitivity to trial products or related products.
* Blood donation except from the donation in this study.
* Subject where it is not possible to obtain sufficient data.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2023-07-04 (Actual); Study Completion 2023-07-04 (Actual)

PRIMARY OUTCOMES:
The change in bone turnover marker CTX. | 1 year
  Changes in fasting blood samples of bone turnover marker CTX attained at randomization, 3 months visit and 12 months visit (final visit)
The change in bone turnover marker P1NP. | 1 year
  Changes in fasting blood samples of bone turnover marker (P1NP) attained at randomization, 3 months visit and 12 months visit (final visit)
The change in loss of bone mineral density. | 1 year
  Changes in DXA scan results of BMD (femur) and BMD (lumbar spine) attained at randomization and 12 months visit (final visit)

SECONDARY OUTCOMES:
Changes in blood parameters of iPTH | 1 year
  Changes in fasting blood samples of iPTH attained at randomization and 12 months visit (final visit)
Changes in blood parameters of Vitamin D | 1 year
  Changes in fasting blood samples of vitamin D attained at randomization and 12 months visit (final visit)
Changes in blood parameters of total calcium | 1 year
  Changes in fasting blood samples of total calcium attained at randomization and 12 months visit (final visit)
Changes in blood parameters of phosphate | 1 year
  Changes in fasting blood samples of phosphate attained at randomization and 12 months visit (final visit)

OTHER OUTCOMES:
Changes in BMI | 1 year
  Changes in BMI from randomization to 12 months visit (final visit)
Changes in physical activity | 1 year
  Changes in physical activity level attained by IPAQ from randomization to 12 months visit (final visit)
Changes in habitual dietary intake | 1 year
  Changes in habitual dietary intake attained by Myfood24 7-day recording from randomization to 12 months visit (final visit)
Changes in fecal pH | 1 year
  Changes in fecal pH from randomization to 12 months visit (final visit)
Changes in gut microbiome | 1 year
  Changes in microbial taxonomy and microbial gene content measured via sequencing of DNA extracted from fecal samples from randomization to 12 months visit (final visit)
Changes in urinary metabolites | 1 year
  Changes in urine metabolites from randomization to 12 months visit (final visit) by NMR spectroscopy to detect and quantify about 50 metabolites including creatinine, amines, amino acids, alcohols, carboxylic acids including short-chain fatty acids, keto acids, purine, pyridine and pyrimidine derivatives, sugars and derivatives.
Changes in fecal metabolites | 1 year
  Changes in fecal metabolites from randomization to 12 months visit (final visit) by NMR spectroscopy to detect and quantify about 50 metabolites including creatine, creatinine, amines, amino acids, carboxylic acids including short-chain fatty acids, keto acids, nucleotides and derivatives.

CONTACTS AND LOCATIONS:
Overall Officials: Mette F Hitz, Doctor, Principal Investigator — Zealand University Hospital, Køge
Locations (2):
- Denmark (2):
  - Copenhagen University, Department of Nutrition, Exercise and Sports, Section for Clinical and Preventive Nutrition, Copenhagen, Frederiksberg
  - Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No
The results will be analyzed and attempted published in international journals regardsless of whether the study leads to positive, negative or inconclusive results. The study protocol will be registered and made publicly avalailable at www.clinicaltrials.gov.